CLINICAL TRIAL: NCT06122090
Title: Evaluation of Laser-assisted Drug Delivery of Bimatoprost for the Treatment of Hypertrophic Scar Hypopigmentation: A Within Patient-Controlled Trial in Skin of Color
Brief Title: Treatment of Hypopigmented Scars With Bimatoprost
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Latham Fund (Unknown)
Responsible Party: Principal Investigator, Bonnie Carney, Research Scientist, Department of Burn Research, Principal Investigator, Medstar Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00006189
Record Dates: First submitted 2023-08-11; First posted 2023-11-08 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Scars; Hypopigmented Scar; Hypopigmented Skin; Burn Scar; Scarring; Cicatrix, Hypertrophic; Cicatrix; Pigmentation Disorder; Burns Laser
Keywords: burn hypertrophic scar; burn scar hypopigmentation; scar; hypopigmentation; dyschromia; pigmentation abnormality
MeSH Terms: conditions — Cicatrix; Vitiligo; Cicatrix, Hypertrophic; Pigmentation Disorders; Hypopigmentation | interventions — Bimatoprost; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Bimatoprost will be delivered to the scars using laser-assisted drug delivery in this arm
  Interventions: Drug: Bimatoprost
- Control (Sham Comparator): Saline control will be delivered to the scars using laser-assisted drug delivery in this arm
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Bimatoprost — Bimatoprost will be delivered with laser
  Arms: Treatment
Drug: Saline — Saline control will be delivered with laser
  Arms: Control

SUMMARY:
Patients who have hypo-pigmented burn scar will have two scars chosen and randomized to treated scar and control scar. The subject will then have both scars treated with fractional ablative CO2 laser (FLSR). The treated scar will have bimatoprost delivered through the laser channels, while the control will have the vehicle (normal saline) only delivered. The treatment will continue for 14 days with twice daily application. The scars will then be monitored at a 2-week follow-up visit where levels of melanin will be evaluated. Tissue punch biopsies will also be used to evaluate the mechanism of action of bimatoprost. Treatment will occur for 6 sessions at 4-6 week intervals including follow- up visits and evaluations.

DETAILED DESCRIPTION:
If the subject agrees to take part in this study, the subject's scars will be looked at and the investigators will pick two sites that will be involved in the research. Each scar will be "randomized" into one of two study groups. One scar will be the treatment group which will be treated with standard of care therapies plus the fractionated ablative CO2 laser and topical bimatoprost drug. The other scar will be the control group which will be treated with standard of care therapies, the fractional ablative CO2 laser, and a control solution. Randomization means that either of the two scars has an equal chance of being designated as the treatment or control group. It is like flipping a coin. Neither the subject nor the investigators will choose what scar will be treated or control. Each half has a 50% chance of being placed in either group.

This study will take place in an outpatient setting. Subjects will not be admitted to the hospital overnight. Patients who enter the study will need to be able to follow up for regular appointments with the burn department.

Before the investigators start the laser treatment, the subject will come in for a pre-treatment visit where the investigators will collect information about the scars such as pictures, non-invasive probes, non-invasive imaging (ultrasound), and questionnaires filled out by the subject and the provider. These questionnaires will be related to the symptoms and appearance of scars. The questionnaires will also evaluate overall psychological health. There will also be a blood draw where less than 2 tablespoons of blood are collected. It is estimated this visit will take less than 1 hour. The investigators will also collect information from the medical record about prior surgical and medical history.

Laser treatments will occur at approximately 4-8-week intervals depending on what the Burn Center scheduling department allows. For completion of this study, the subject will undergo 6 laser treatments which should take about 6-12 months. During each laser treatment visit, the treated scar will have the drug (bimatoprost) rubbed on top of the scar while the subject is having their surgery. The subject will then continue to apply these drops to their scar for 14 days after the surgery, once in the morning and once at night. The drug will come in a bottle with a dropper top which the subject will apply a couple of drops to their scar and rub it in. The investigators will tell the subject how much drug to apply based on the size of their scar. This drug will be provided to the subject by the research pharmacy and will not be billed to the subject's insurance. The study team will call to remind the subject about their laser visits and to make sure they are applying the ointment for 14 days. The subject will apply the study drug to one scar and the control drug to the other scar. The investigators will label the containers so subjects will know which one to apply where. The subject will write down when they apply their medications in a diary entry that will be completed daily for 14 days after each laser procedures.

While most patients with burn scars undergo 6 treatments, and this is the goal for this study, sometimes depending on how the subject's scar is responding to treatment, they along with their clinical team may decide to stop treatments before the subject gets to 6 treatments, or continue after 6 treatments. Treatments of scars will stop when the clinical team elects to stop laser treatment.

If this means that the subject will only receive 1, 2, 3, 4, or 5 laser treatments instead of 6, then the subject will go into long-term follow up for the study. However, if that means the subject will get more than 6 laser treatments as a part of their clinical care, they will no longer apply the investigational drug after 6 treatments. The subject's laser surgeries will not be any longer because of their participation in the study, they will take the same amount of time as if they were not a study participant.

Treated scars will be assessed at these regular intervals: within 18 days ± 3 days following each treatment, and 12 months ± 1 month after the final study laser treatment. During the 12-month follow-up, there will also be a blood draw where less than 2 tablespoons of blood are collected. The study team will call the subject to remind them about their follow-up visits so that they can make every effort to be there. The follow-up visits will take about 30 minutes-1 hour and will be with a member of the research team. These visits can be scheduled right after the subject will be returning to see their rehab therapist for their post-laser assessment. The subject would have to come back to these follow-ups as a part of their routine clinical care any way if they were not a part of this research study.

A 3mm punch biopsy will be collected from the treatment and control scars at each laser treatment visit (Laser surgery #1, #2, #3, #4, #5, and #6). Two 3mm punch biopsies will be taken of non-burned skin only at the first laser treatment. These biopsies will be taken when the subject is under anesthesia as a part of their laser surgery.

At study entrance and at each study visit, photographs will be taken of the control and treated scars. All photographs taken for the purpose of this study will be taken by a study camera, with images stored on a password-protected secure server. These photographs will be labeled with a study ID number. All efforts will be made to minimize the amount of identifiable information such as the face or tattoos in these photos.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years
2. Cutaneous trauma resulting in hypopigmented scar
3. 2 different hypopigmented scars (at least 30cm2 each) with at least 2 inches of normal skin, hyperpigmented scar, or hypopigmented scar separating each hypopigmented study site scar

Exclusion Criteria

1. Target hypopigmented scar to face or genitalia
2. Known allergy to bimatoprost
3. Known allergy to lidocaine
4. Positive urine pregnancy test in women of childbearing potential (per point of care test)
5. Lactating women (self-reported)
6. Prisoner status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Area of pigmentation | follow-up number 6, an average of 8 months
  area of pigmentation within control and treated scars

SECONDARY OUTCOMES:
Melanin Index | follow-up number 6, an average of 8 months
  Melanin index of hypopigmented burn scars (minimum=500, maximum=950, higher score correlates with a better outcome)
Differential gene expression of tyrosinase | follow-up number 6, an average of 8 months
  pigmentation signaling molecules within tissue punch biopsies
Differential gene expression of tyrosinase-related protein 1 | follow-up number 6, an average of 8 months
  pigmentation signaling molecules within tissue punch biopsies
Differential gene expression of tyrosinase-related protein 2 | follow-up number 6, an average of 8 months
  pigmentation signaling molecules within tissue punch biopsies

OTHER OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) | follow-up number 6, an average of 8 months
  minimum=0, maximum=10, higher score correlates with worse outcomes
VanCouver Scar Scale | follow-up number 6, an average of 8 months
  minimum=0, maximum=13, higher score correlates with worse outcomes
Non-invasive measurement of melanin | follow-up number 6, an average of 8 months
  melanin index value will be obtained using the Delfin Technologies SkinColorCatch Probe
Non-invasive measurement of elasticity | follow-up number 6, an average of 8 months
  instant skin elasticity value will be obtained using the Delfin Technologies Elastimeter Probe
Non-invasive measurement of stiffness | follow-up number 6, an average of 8 months
  stiffness (N/m) value will be obtained using the Checkline Durometer

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States